CLINICAL TRIAL: NCT07068295
Title: A Study Investigating the Pharmacokinetic and Pharmacodynamic Properties and Safety and Tolerability of NNC0471-0119 H When Administered as Bolus in a Continuous Subcutaneous Insulin Infusion Regimen in Participants With Type 2 Diabetes
Brief Title: A Study to Test How Insulin NNC0471-0119 H Works in the Body in Participants With Type 2 Diabetes When Given by an Insulin Pump
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN1471-5026; U1111-1283-0507 (Other: World Health Organization (WHO)); 2024-520230-29 (Other: European Medical Agency (EMA))
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NNC0471-0119 H then Insulin Aspart (Experimental): Participants will receive NNC0471-0119 H subcutaneously (s.c.) in period 1 followed by insulin aspart s.c. in period 2.
  Interventions: Drug: NNC0471-0119 H; Drug: Insulin Aspart
- Insulin Aspart then NNC0471-0119 H (Active Comparator): Participants will receive insulin aspart s.c. in period 1 followed by s.c. NNC0471-0119 H in period 2.
  Interventions: Drug: NNC0471-0119 H; Drug: Insulin Aspart

INTERVENTIONS:
Drug: NNC0471-0119 H — NNC0471-0119 H will be administered subcutaneously.
Drug: Insulin Aspart — Insulin aspart will be administered subcutaneously.

SUMMARY:
This study looks at the effect and safety of a new fast-acting insulin (NNC0471-0119) in people with type 2 diabetes when given by an insulin pump. The study tests how fast insulin NNC0471-0119 enters bloodstream, how long it stays there and how much it lowers blood sugar. The new insulin NNC0471-0119 will be compared to insulin aspart. The study will last for about 13-67 days (or a half to 2 months).

ELIGIBILITY:
Inclusion Criteria:

* Male or female (sex at birth).
* Age 18-69 years (both inclusive) at the time of signing the informed consent.
* Diagnosed with Type 2 Diabetes (T2D) greater than or equal to (≥) 180 days before screening.
* Treated with any injectable insulin, except once-weekly insulin, ≥ 180 days before screening.
* Current daily insulin treatment between 0.2 and 1.2 Insulin units per kilogram per day [(I) U/kg/day] (both inclusive) with or without the following anti-diabetic drugs with stable doses ≥ 90 days prior to the day of screening:
* Any metformin formulation
* Dipeptidyl peptidase-4 inhibitor (DPP4i)
* Sodium-glucose Cotransporter-2 inhibitor (SGLT2i)
* Body mass index (BMI) between 18.5 and 34.9 kg/m2 (both inclusive) at screening.
* HbA1c lesser than or equal to (≤) 9.5%

Exclusion Criteria:

* Known or suspected hypersensitivity to study intervention(s) or related products.
* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using adequate contraceptive methods.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2026-01-12 (Estimated); Study Completion 2026-01-12 (Estimated)

PRIMARY OUTCOMES:
AUC(GIR,0-1h,basal-corrected): Area under the basal-corrected glucose infusion rate (GIR)-time curve from 0 to 1 hour | 0 to 1 hour after bolus infusion
  Measured in milligram per kilogram (mg/kg).

SECONDARY OUTCOMES:
AUC(GIR,0-t,basal-corrected): Area under the basal-corrected GIR-time curve from 0 to t | 0 to 11 hours after bolus infusion
  Measured in mg/kg.
AUC(GIR,0-1h,basal-corrected)/AUC(GIR,0-t,basal-corrected): Ratio of the area under the basal-corrected GIR-time curve from 0 to 1 hour and 0 to t | 0 to 11 hours after bolus infusion
  Measured in percentage (%).
GIR (max,basal-corrected): Maximum observed basal-corrected GIR | 0 to 11 hours after bolus infusion
  Measured in milligrams per (kilogram *minute) (mg/[kg*min]).
AUC(NNC0471-0119,0-30min,basal-corrected)/AUC (NNC0471-0119,0-t,basal-corrected): Ratio of the basal-corrected area under the serum NNC0471-0119 concentration time curve from 0 to 30 minutes and 0 to t | 0 to 11 hours after bolus infusion
  Measured in %.
AUC(NNC0471-0119,0-t,basal-corrected): Area under the basal-corrected serum NNC0471-0119 concentration time curve from 0 to t | 0 to 11 hours after bolus infusion
  Measured in hours*picomole per liter (h*pmol/L).
AUC(NNC0471-0119,0-30min,basal-corrected): Area under the basal-corrected serum NNC0471-0119 concentration time curve from 0 to 30 minutes | 0 to 30 minutes after bolus infusion
  Measured in h*pmol/L.
AUC(NNC0471-0119,2h-t,basal-corrected): Area under the basal-corrected serum NNC0471-0119 concentration time curve from 2 hours to t | 2 to 11 hours after bolus infusion
  Measured in h*pmol/L.
AUC(NNC0471-0119,2h-t,basal-corrected)/AUC(NNC0471-0119 H,0-t,basal-corrected): Ratio of the basal-corrected area under the serum NNC0471-0119 concentration time curve from 2 hours to t and 0 to t | 0 to 11 hours after bolus infusion
  Measured in %.
C(max,NNC0471-0119,basal-corrected): Maximum observed basal-corrected serum NNC0471-0119 concentration | 0 to 11 hours after bolus infusion
  Measured in picomoles per litre (pmol/L).
t(early50%Cmax,NNC0471-0119,basal-corrected): Time to early 50% maximum observed basal-corrected serum NNC0471-0119 concentration | 0 to 11 hours after bolus infusion
  Measured in minutes (Min).
t(late50%Cmax,NNC0471-0119,basal-corrected): Time to late 50% maximum observed basal-corrected serum NNC0471-0119 concentration | 0 to 11 hours after bolus infusion
  Measured in min.
Number of adverse events (AEs) | From start of first investigational medicinal product (IMP) basal rate infusion (day -1) until completion of post-treatment end of study visit (up to 67 days)
  Measure in number of events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com